CLINICAL TRIAL: NCT03658057
Title: Recording Sympathetic Nerve Activity From the Skin During Surgery Under General Anesthesia : a Pilot Study
Brief Title: Measurement of the Skin Sympathetic Nerve Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: SKNA pilot
Record Dates: First submitted 2018-08-29; First posted 2018-09-05 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Skin Sympathetic Nerve Activity During General Anesthesia in Patients Undergoing Breast Cancer Surgery
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ROC (Active Comparator): Neuromuscular blockade is performed in the ROC group by administering rocuronium 0.4~0.8mg/kg before the insertion of laryngeal airway.
  Interventions: Drug: Rocuronium
- Control (No Intervention): Neuromuscular blockade is not performed.

INTERVENTIONS:
Drug: Rocuronium — whether neuromuscular blockade by administering rocuronium is performed or not.
  Arms: ROC

SUMMARY:
Sympathetic nerve activity can be measured transcutaneously in awake patients by computer-based filtering of raw signal obtained via skin leads attached on the chest. Electrocardiogram can be removed by applying a high-pass filter setting of 150 Hz. Electromyogram can be filtered by applying a high-pass filter setting of 500 Hz or a band-pass filter setting of 500-1000 Hz.

However, it is not known whether the skin sympathetic nerve activity (SKNA) can be measured in anesthetized and/or paralyzed patients. Therefore, we planned this pilot study to observe whether the SKNA can be obtained in these patients. If the SKNA ca be observed, it will be presented in milivolt (uV).

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled to undergo resection of breast cancer under general anesthesia after insertion of laryngeal mask airway

Exclusion Criteria:

* Autonomic nervous system disease
* Medication acting on the autonomic nervous system
* Refuse to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-08-31 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The skin sympathetic nerve activity presented as uV obtained via skin leads. | During surgery/anesthesia
  A few studies reported that skin sympathetic nerve activity (SKNA) signal could be potentially observed by applying a high-pass filter of 500 Hz or a band-pass filter of 500~1000 Hz to electric signal from skin leads attached on the skin of the chest in awake volunteers. However, it is not known if it would be also possible to observe the SKNA signal in anesthetized patients. Also, there is no established method for quantitative or qualitative assessment of the SKNA signal.

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, Jeon, Study Director — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea